CLINICAL TRIAL: NCT03427333
Title: Rook Epicardial Access Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Talon Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: M064-035
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Ventricular Tachycardia; Arrythmia
Keywords: VT; Pacemaker Lead Extraction; epicardial access; pericardial access
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Intervention Model: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- The Rook® Epicardial Access Kit (Experimental): The Rook® Epicardial Access Kit will be used to gain access the epicardial surface of the heart via a subxiphoid approach in adult patients with a normal, non-distended pericardial space.
  Interventions: Device: The Rook® Epicardial Access Kit

INTERVENTIONS:
Device: The Rook® Epicardial Access Kit — Use of the Rook Epicardial Access Kit to gain access to the normal, non distended pericardial space.

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of the Talon Surgical Rook® Epicardial Access Kit as a pericardial access device. The Rook® Epicardial Access Kit will be used to gain access the epicardial surface of the heart via a subxiphoid approach in adult patients with a normal, non-distended pericardial space.

DETAILED DESCRIPTION:
This is a first-in-human, prospective, non-randomized, single arm study to confirm the efficacy and safety of the Talon Surgical Rook® Epicardial Access Kit to achieve guidewire access to the pericardial space. Patients who are clinically indicated to undergo a procedure that requires percutaneous access to the normal, non-distended, pericardial space will be considered for enrollment into this clinical trial. This may include, but is not limited to, patients who require pericardial access for epicardial ablation procedure or for pigtail catheter placement during pacemaker lead extraction. The study population will consist of both male and female patients of at least 18 years of age. In addition, eligible patients will have a life expectancy of at least 6 months based on a physician's assessment of the patient's medical condition. Patients who meet all inclusion and non-exclusion criteria, who are willing to comply with study follow-up requirements, and for whom documented informed consent is obtained, will be eligible for enrollment in the study. Enrollment occurs when the device enters the body.

Patients who undergo attempted use of a study device (patient leaves procedure room with device having entered the body at some point during the procedure), regardless of whether or not the device was successfully used for pericardial access, will be followed through discharge or up to 4 days post procedure, whichever comes first.

The study will include a minimum of 10 patients and up to 30 patients with the study devices used for pericardial access. Multiple study site may be utilized. The duration of participation for each enrolled patient who utilizes a study device for pericardial access will be through hospital discharge, or up to 4 days post procedure, whichever comes first.

A study physician will utilize the Rook® Epicardial Access Kit to gain access to the pericardial space. The physician will follow the patient through hospital discharge, or up to 4 days post procedure, whichever comes first, for adverse events, and other device or procedure related observations. The study coordinator or designated study personnel at the Principle Investigator's office will be responsible for collecting data from the procedure and hospital stay which will be necessary for completion of case report form for the index procedure and subsequent follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is clinically indicated to undergo a procedure that requires percutaneous access to the normal, non-distended, pericardial space.
* Patient is willing and able to provide written informed consent.

Exclusion Criteria:

* Subject is younger than 18 years of age
* Previous cardiac surgery
* Myocardial infarction within 4 weeks prior to procedure
* Class IV NYHA (New York Heart Association) heart failure symptoms
* Subject with an active systemic infection
* Known carotid artery stenosis greater than 80%
* Presence of thrombus in the left atrium
* Congenital absence of a pericardium
* Coagulopathy
* Hemodynamic Instability
* Acute conditions (i.e. electrolyte abnormality, acute ischemia, drug toxicity)
* Severe hepatic dysfunction or enlargement
* Subject has Body Mass Index > 40
* Life expectancy less than 6 months
* Subject is pregnant
* Subject is currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study
* Subject has known or suspected allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Patient in Whom Successful Pericardial Access was Achieved Through Use of the Rook Epicardial Access Kit | At time of intervention.
  Standard x-ray (fluoroscopy) will be used to confirm that the Talon Surgical Rook® Epicardial Access Kit facilitated successful placement of a guidewireinto the pericardial space. Successful placement of the guidewire into the pericardial space will be noted for each patient. The percentage of patients in whom pericardial access was successful will be reported.

SECONDARY OUTCOMES:
Number of Participants with Device or Procedure Related Adverse Events as Adjudicated by the Clinical Event Committee | Up to 4 days post procedure.
  Occurrence of CEC-adjudicated device or procedure related adverse events through hospital discharge or up to 4 days post procedure, whichever comes first, will be documented for each patient. The total number of patients with adverse events and the number of each adverse events will be reported. This outcome will also be reported as a percentage.
Speed of Access | At time of intervention
  Time from skin incision to confirmed guidewire access to the pericardial space.
Ease of Use | At time of intervention.
  Evaluation of the study procedure compared to the standard of care pericardial access procedure with a Tuohy Needle by clinician survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czechia